CLINICAL TRIAL: NCT00714311
Title: A Randomized-Controlled Trial of Transference-Focused Psychotherapy vs. Treatment by Experienced Community Psychotherapists for Borderline Personality Disorder
Brief Title: Efficacy of Transference-Focused Psychotherapy for Borderline Personality Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Responsible Party: Principal Investigator, doerings, Univ.-Prof. Dr. med., University Hospital Muenster
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1106/04; 10636; DPG0802
Record Dates: First submitted 2008-07-09; First posted 2008-07-14 (Estimated); Results first posted 2015-02-16 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-02

CONDITIONS: Borderline Personality Disorder
Keywords: borderline personality disorder; randomized controlled trial; Transference-Focused Psychotherapy; treatment by experienced community psychotherapists
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TFP (Active Comparator): Transference-Focused Psychotherapy
  Interventions: Behavioral: Transference-Focused Psychotherapy
- ECP (Active Comparator): treatment by experienced community psychotherapists
  Interventions: Behavioral: treatment by experienced community psychotherapists

INTERVENTIONS:
Behavioral: Transference-Focused Psychotherapy — Outpatient psychotherapy according to the treatment manual, sessions of 50 minutes twice per week
  Arms: TFP
Behavioral: treatment by experienced community psychotherapists — Outpatient psychotherapy in private practices or outpatient units of psychiatric hospitals. Licensed psychotherapists with experience and special interest in the treatment of borderline patients are treating according to the method they have learned.
  Arms: ECP

SUMMARY:
The purpose of this study is to find out whether Transference-Focused Psychotherapy (TFP) is effective in the treatment of Borderline Personality Disorder.

DETAILED DESCRIPTION:
Borderline personality disorder represents a sever clinical condition that affects 1-2% of the community and is characterized by a pervasive instability of interpersonal relationships, self-image, and affects, as well as a marked impulsivity; up to 10% of the patients commit suicide.

Transference-Focused Psychotherapy (TFP) is one psychotherapeutic approach among five that have been manualized and evaluated in RCTs. So far, TFP has not been compared to a control condition which is a crucial step in the evaluation of the efficacy of a psychosocial intervention.

This study is an RCT that compares one year of outpatient TFP to treatment by experienced community psychotherapists for borderline personality disorder.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent to the participation in the study
* Diagnosis of BPD according to DSM-IV as assessed using the SCID-II
* Age between 18 and 45 years
* Sufficient knowledge of the German language

Exclusion Criteria:

* Diagnosis of schizophrenia, bipolar disorder, severe substance abuse, organic pathology, or mental retardation according to DSM-IV as assessed using the SCID-I
* Diagnosis of antisocial personality disorder according to DSM-IV as assessed using the SCID-II

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2004-10; Primary Completion 2009-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Doering, MD, Principal Investigator — University of Muenster, Germany
Locations (2):
- Dept. of Psychoanalysis and Psychotherapy, Medical University Vienna, Vienna, Vienna, Austria
- Dept. of Psychiatry, Technical University of Munich, Munich, Bavaria, Germany

REFERENCES:
- [Background] Clarkin JF, Levy KN, Lenzenweger MF, Kernberg OF. Evaluating three treatments for borderline personality disorder: a multiwave study. Am J Psychiatry. 2007 Jun;164(6):922-8. doi: 10.1176/ajp.2007.164.6.922. PMID 17541052
- [Background] Levy KN, Meehan KB, Kelly KM, Reynoso JS, Weber M, Clarkin JF, Kernberg OF. Change in attachment patterns and reflective function in a randomized control trial of transference-focused psychotherapy for borderline personality disorder. J Consult Clin Psychol. 2006 Dec;74(6):1027-1040. doi: 10.1037/0022-006X.74.6.1027. PMID 17154733
- [Background] Kernberg OF, Yeomans FE, Clarkin JF, Levy KN. Transference focused psychotherapy: overview and update. Int J Psychoanal. 2008 Jun;89(3):601-20. doi: 10.1111/j.1745-8315.2008.00046.x. PMID 18558958
- [Derived] Schmitz-Riol S, Fuchshuber J, Herpertz J, Buchheim A, Horz-Sagstetter S, Rentrop M, Fischer-Kern M, Buchheim P, Taylor J, Tmej A, Weihs KL, Lane RD, Doering S. Emotion word repertoire in the adult attachment interview predicts a reduction of non-suicidal self-injury in the psychotherapy of borderline personality disorder. BMC Psychiatry. 2025 Aug 28;25(1):832. doi: 10.1186/s12888-025-07300-6. PMID 40877786
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617
- [Derived] Storebo OJ, Stoffers-Winterling JM, Vollm BA, Kongerslev MT, Mattivi JT, Jorgensen MS, Faltinsen E, Todorovac A, Sales CP, Callesen HE, Lieb K, Simonsen E. Psychological therapies for people with borderline personality disorder. Cochrane Database Syst Rev. 2020 May 4;5(5):CD012955. doi: 10.1002/14651858.CD012955.pub2. PMID 32368793
- [Derived] Doering S, Horz S, Rentrop M, Fischer-Kern M, Schuster P, Benecke C, Buchheim A, Martius P, Buchheim P. Transference-focused psychotherapy v. treatment by community psychotherapists for borderline personality disorder: randomised controlled trial. Br J Psychiatry. 2010 May;196(5):389-95. doi: 10.1192/bjp.bp.109.070177. PMID 20435966

RESULTS

PARTICIPANT FLOW:
Groups:
- Transferenced-Focused Psychotherapy: Transferenced-Focused Psychotherapy (TFP)
- Experienced Community Psychotherapists: Experienced Community Psychotherapists (ECP)
Period: Overall Study
Arm/Group | Transferenced-Focused Psychotherapy | Experienced Community Psychotherapists
Started | 52 | 52
Completed | 39 | 30
Not Completed | 13 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Transferenced-Focused Psychotherapy | Experienced Community Psychotherapists | Total
Number analyzed (Participants) | 52 | 52 | 104
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 52 | 52 | 104
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.46 (6.8) | 27.19 (7.5) | 27.33 (7.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 52 | 104
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Austria | 20 | 20 | 40
  Germany | 32 | 32 | 64

OUTCOME MEASURES:

1. Primary Outcome: Drop-out
Description: Did not finish one year of treatment.
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Transferenced-Focused Psychotherapy | Experienced Community Psychotherapists
Number analyzed (Participants) | 39 | 30
participants | 13 | 20

2. Primary Outcome: Suicidality (Suicide Attempts)
Time Frame: 1 year
Reporting Status: Not Posted

3. Secondary Outcome: Psychosocial Functioning (Global Assessment of Functioning, GAF-Score)
Time Frame: 1 year
Reporting Status: Not Posted

4. Secondary Outcome: Level of Personality Organization (Structured Interview for Personality Organization, STIPO)
Time Frame: 1 year
Reporting Status: Not Posted

5. Secondary Outcome: Number of Self-harming Acts
Time Frame: 1 year
Reporting Status: Not Posted

6. Secondary Outcome: Self-assessment of Psychopathology (BDI, STAI, BSI)
Time Frame: 1 year
Reporting Status: Not Posted

7. Secondary Outcome: Attachment Style and Reflective Function (Adult Attachment Interview, AAI)
Time Frame: 1 year
Reporting Status: Not Posted

8. Secondary Outcome: Borderline Symptomatology (DSM-IV Criteria)
Time Frame: 1 month
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- Transference-Focused Psychotherapy: Transference-Focused Psychotherapy (TFP)
  Transference-Focused Psychotherapy: Outpatient psychotherapy according to the treatment manual, sessions of 50 minutes twice per week
- Treatment by Experienced Community Psychotherapists: treatment by experienced community psychotherapists (ECP)
  treatment by experienced community psychotherapists: Outpatient psychotherapy in private practices or outpatient units of psychiatric hospitals. Licensed psychotherapists with experience and special interest in the treatment of borderline patients are treating according to the method they have learned.
Arm/Group | Transference-Focused Psychotherapy | Treatment by Experienced Community Psychotherapists
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes